CLINICAL TRIAL: NCT04236947
Title: Randomized Control Trial of the Effectiveness of the Social Competence Promotion Program for Young Adolescents Aimed at Preventing Substance Use Among Students in Chile
Brief Title: Effectiveness of the Social Competence Promotion Program for Young Adolescents for Substance Use Prevention in Chile
Acronym: SCPP-YA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de los Andes, Chile (Other)
Collaborators: Comisión Nacional de Investigación Científica y Tecnológica (Other Government); University of Talca (Other)
Responsible Party: Principal Investigator, Jorge Gaete, Associate Professor, Universidad de los Andes, Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FONIS SA19I0115
Record Dates: First submitted 2020-01-17; First posted 2020-01-22 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Substance Use
Keywords: Adolescents; Prevention; School; Social Competence Promotion Program for Young Adolescents
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: This study is a randomized control trial with two arms.
Who Masked: Outcomes Assessor
Masking Description: During the assessments, research assistants will be blind to the allocation of schools.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCPP-YA group (Experimental): SCPP-YA adapted to Chile consist of ten sessions promoting self-regulation strategies, prosocial, and problem-solving skills. It also includes a module (6 sessions) specially designed for substance use prevention, developing social competence, and assertiveness to deal with peer pressure. These 16 sessions will be implemented during an academic year (2020), and complemented with three booster sessions the following year (2021).
  Interventions: Behavioral: SCPP-YA
- Control Group (No Intervention): The control schools will continue providing their traditional preventive actions.

INTERVENTIONS:
Behavioral: SCPP-YA — SCPP-YA includes two modules. In the first module of ten sessions, students will learn to employ a 6-step social information processing framework for solving a wide range of real-life problems. The six-step process consists of 1) stop, clam down, and think before you act; 2) say the problem and how you feel; 3) set a positive goal; 4) think of many solutions; 5) think ahead to the consequences and 6) go ahead and try the best plan. The second module offers 1) current and accurate information about the health, social, and legal consequences of substance use, 2) correct mistaken beliefs that students have about substance use, 3) enhances awareness of social and media influences; and 4) teachers assertiveness and critical thinking skills to resist peer pressure.
  Other Names: Social Competence Promotion Program for Young Adolescents; New Haven Program; Mi Mejor Plan
  Arms: SCPP-YA group

SUMMARY:
Substance use has become a significant public health problem, given its magnitude and the treatment gap encountered when a dependency disorder has already been installed. Still, to date, there are no studies in Chile that show the effectiveness of a universal preventive program implemented in educational settings, using a randomized controlled clinical trial design.

This study consists of evaluating the effectiveness of the Social Competence Promotion Program among Young Adolescents (SCPP-YA), which aims to postpone the onset of substance use and reduce their consumption.

This is a randomized controlled clinical trial with two arms, including students of 6th grade from high socioeconomic vulnerability schools in Santiago. The primary outcome is the incidence of tobacco consumption in the last month.

The SCPP-YA consists of 16 sessions that will be implemented during the academic year (2020) and complemented with three booster sessions the following year (2021). This intervention mainly provides strategies for self-regulation, problem-solving, and substance use prevention.

The investigators expect that students in the intervention group will delay the onset of any substance use, especially tobacco, alcohol, and marijuana when compared with students in the control group.

DETAILED DESCRIPTION:
Chilean adolescents face problems in their mental health and risk behaviors, which compromise their development. Among these behaviors, substance use has become a significant public health problem, given its magnitude and the treatment gap encountered when a dependency disorder has already been installed. In Chile, both prevention and treatment were among the Sanitary Aims of the 2010-2020 decade. For many years, different governmental and non-governmental institutions have implemented preventive initiatives in the school population. Still, to date, there are no studies in Chile that show the effectiveness of a universal preventive program implemented in educational settings, using a randomized controlled clinical trial design.

This study consists of evaluating the effectiveness of the Social Competence Promotion Program among Young Adolescents (SCPP-YA), which aims to postpone the onset of substance use and reduce their consumption.

This is a randomized controlled clinical trial with two arms, including students of 6th grade from high socioeconomic vulnerability schools in Santiago. Ten schools will be randomly allocated to the intervention group and the control group in a 1:1 ratio. Assessments of students will be carried out at baseline, post-intervention, and 12 months after the end of the intervention. The primary outcome is the incidence of tobacco consumption in the last month. The SCPP-YA consists of 10 student sessions providing self-regulation strategies, promotion of prosocial skills, and a method of problem-solving. Additionally, it includes a 6-session module specially designed for substance use prevention. These 16 sessions will be implemented during the academic year (2020) and complemented with three booster sessions the following year (2021).

The investigators expect that students in the intervention group will delay the onset of any substance use, especially tobacco, alcohol, and marijuana when compared with students in the control group.

ELIGIBILITY:
Inclusion Criteria:

1. Schools having primary education (Year 1 to Year 8)
2. Schools located in Santiago (Chile)
3. Schools having a vulnerability index (School Vulnerability Index - National System of Equality Allocation (IVE-SINAE)) ≥ 50%*
4. Mixed-sex schools.
5. Schools willing to participate under the conditions of the study before randomization.

   * The IVE-SINAE is built taking into account several students' and parental variables: health, family income, receiving state benefits. This percentage means the proportion of students in a school who are in most need.

Exclusion Criteria:

1. Schools that are implementing other substance use prevention program similar to the contents and methodology of "Mi Mejor Plan" targeting the same grade.

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Cigarette use in the last month | Past 30-day period
  Measured with the European Drug Addiction Prevention Trial Questionnaire (EU-Dap) validated in Chile. Students will be asked: How many times participants have smoked cigarettes in the last 30 days

SECONDARY OUTCOMES:
Alcohol use in the last month | Past 30-day period
  Measured with the European Drug Addiction Prevention Trial Questionnaire (EU-Dap) validated in Chile. Students will be asked: How many times participants have drink alcohol beverages in the last 30 days
Marijuana use in the last month | Past 30-day period
  Measured with the European Drug Addiction Prevention Trial Questionnaire (EU-Dap) validated in Chile. Students will be asked: How many times participants have consumed marijuana in the last 30 days
Social problem-solving | Last 3 months
  Measured with Social Problem-Solving Inventory, short version. This is a 25-item instrument that measures several problem-solving skills.
Emotional regulation | Last 3 months
  Measured with Emotion Regulation Questionnaire for Children and Adolescents (ERQ-CA).This is a 10-item instrument that measures emotional regulation.
Socio-emotional skills | Last 3 months
  Measured with Strengths and Difficulties Questionnaire (SDQ). This is a 25-item instrument that measures emotional, conduct, peer and hyperactivity/inattention problems
Sense of school membership | Last 3 months
  Measured with the Psychological Sense of School Membership scale (PSSM). This is a scale with 13 items that refers to the student's perceptions of the respect and acceptance that teachers and other students show him or her, as well as his or her sense of belonging.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de los Andes, Santiago, Chile

IPD SHARING:
Plan to Share IPD: Undecided
The investigators plan to share data using "UK Data Service". The investigators will never compromise participant privacy, neither schools nor students.

REFERENCES:
- [Derived] Ramirez S, Rios N, Rojas-Barahona CA, Carcamo M, Sepulveda-Panaloza A, Araya R, Gaete J. Acceptability, feasibility, fidelity and quality implementation of the culturally adapted version of the Social Competence Promotion Program among Young Adolescents ("Mi Mejor Plan") to prevent substance use among adolescents in Chile: a pilot randomized control study. BMC Public Health. 2025 May 20;25(1):1860. doi: 10.1186/s12889-025-23033-3. PMID 40394545
- [Derived] Gaete J, Inzunza C, Ramirez S, Valenzuela D, Rojas C, Araya R. The Social Competence Promotion Program among Young Adolescents (SCPP-YA) in Chile ("Mi Mejor Plan") for substance use prevention among early adolescents: study protocol for a randomized controlled trial. Trials. 2022 Jun 30;23(1):542. doi: 10.1186/s13063-022-06472-w. PMID 35773714